CLINICAL TRIAL: NCT02785354
Title: Engel 2: REal-life aNticoaGulants Comparative bEnefit-risk in Nonvalvular Atrial fibrilLation (NVAF) in France
Brief Title: Anticoagulants Comparative Benefit-risk Ratio in Real Life
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.263
Record Dates: First submitted 2016-05-25; First posted 2016-05-27 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- NOAC: New oral anticoagulant groups
- VKA: VKA group

SUMMARY:
The study is an analysis using the French national health insurance database, six months after the beginning of NOAC launch in the NVAF indication.

The aim is to compare the one-year, two-year and three-year benefit-risk (major bleeding, arterial thrombotic events, myocardial infarction (MI), death) between patients starting a NOAC and patients starting a VKA for NVAF in 2013

ELIGIBILITY:
Inclusion criteria:

Patients with NVAF with a first reimbursed dispensation of Pradaxa®, Xarelto®, or VKA in 2013, with no other identified indication for anticoagulation; Without any VKA or NOAC (Pradaxa®, Xarelto®, or Eliquis®) reimbursed dispensation for the last 3 years before the first reimbursed dispensation of Pradaxa®, Xarelto®, or VKA

Exclusion criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New users of NOAC or VKA for NVAF
Sampling Method: Non-Probability Sample
Enrollment: 103101 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2016-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.263.1 Boehringer Ingelheim Investigational Site, Multiple Locations, France

REFERENCES:
- [Derived] Blin P, Dureau-Pournin C, Benichou J, Cottin Y, Mismetti P, Abouelfath A, Lassalle R, Droz C, Moore N. Comparative Real-Life Effectiveness and Safety of Dabigatran or Rivaroxaban vs. Vitamin K Antagonists: A High-Dimensional Propensity Score Matched New Users Cohort Study in the French National Healthcare Data System SNDS. Am J Cardiovasc Drugs. 2020 Feb;20(1):81-103. doi: 10.1007/s40256-019-00359-z. PMID 31254174
- [Derived] Blin P, Dureau-Pournin C, Cottin Y, Benichou J, Mismetti P, Abouelfath A, Lassalle R, Droz C, Moore N. Comparative Effectiveness and Safety of Standard or Reduced Dose Dabigatran vs. Rivaroxaban in Nonvalvular Atrial Fibrillation. Clin Pharmacol Ther. 2019 Jun;105(6):1439-1455. doi: 10.1002/cpt.1318. Epub 2019 Feb 6. PMID 30499605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study ENGEL 2 is a real-world historical cohort study in the French nationwide healthcare claims and hospitalization database (SNIIRAM) including new users of DOAC or VKA for nonvalvular atrial fibrillation (NVAF) in 2013 with a follow-up for one year (main objective).
Pre-assignment Details: The main objective was to compare the risk & effectiveness for dabigatran vs VKA, & for rivaroxaban vs VKA. The main analysis was done for hdPS matched patients (pts.) with atrial fibrillation (AF) diagnosis information in the database.
Groups:
- Dabigatran: Patients with a first dispensing of dabigatran in 2013 for NVAF.
- Rivaroxaban: Patients with a first dispensing of rivaroxaban in 2013 for NVAF.
- Vitamin K Antagonists: Patients with a first dispensing of VKA in 2013 for NVAF.
Period: Overall Study
Arm/Group | Dabigatran | Rivaroxaban | Vitamin K Antagonists
Started | 27060 | 31388 | 44653
Completed | 27060 | 31388 | 44653
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The main analysis was on matched patients 1:1 on the date of the first drug (DOAC or VKA) dispensing (± 2 weeks), gender, age at index date (± 1 year) and hdPS (± 0.05).Baseline measures were presented for overall treatment groups and matched populations: dabigatran vs VKA and rivaroxaban vs VKA.
Groups:
- Dabigatran: Patients with a first dispensing of dabigatran in 2013 for NVAF, matched 1:1 on the date of the first dispensing, gender, age at index date, and hdPS.
- Rivaroxaban: Patients with a first dispensing of rivaroxaban in 2013 for NVAF, matched 1:1 on the date of the first dispensing, gender, age at index date, and hdPS.
- Vitamin K Antagonists: Patients with a first dispensing of VKA in 2013 for NVAF, matched 1:1 on the date of the first dispensing, gender, age at index date, and hdPS.
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Rivaroxaban | Vitamin K Antagonists | Total
Number analyzed (Participants) | 27060 | 31388 | 44653 | 103101
Age, Customized [Mean (Standard Deviation); unit: Years] — Population: The main analysis was on matched patients 1:1 on the date of the first drug (DOAC or VKA) dispensing (± 2 weeks), gender, age at index date (± 1 year) and hdPS (± 0.05).Baseline measures were presented for overall treatment groups and matched populations: dabigatran vs VKA and rivaroxaban vs VKA.
  Years
    Overall | 73.2 (11.8) | 73.2 (11.8) | 77.9 (11.1) | 75.2 (11.7)
    Dabigatran vs VKA (matched pop): number analyzed (Participants) | 20489 | 0 | 20489 | 40978
    Dabigatran vs VKA (matched pop) | 75.3 (10.7) |  | 75.4 (10.7) | 75.4 (10.7)
    Rivaroxaban vs VKA (matched pop): number analyzed (Participants) | 0 | 23053 | 23053 | 46106
    Rivaroxaban vs VKA (matched pop) |  | 75.3 (10.7) | 75.4 (10.7) | 75.4 (10.7)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The main analysis was on matched patients 1:1 on the date of the first drug (DOAC or VKA) dispensing (± 2 weeks), gender, age at index date (± 1 year) and hdPS (± 0.05).Baseline measures were presented for overall treatment groups and matched populations: dabigatran vs VKA and rivaroxaban vs VKA.
  Participants
    Overall: Male | 15253 | 17653 | 22868 | 55774
    Overall: Female | 11807 | 13735 | 21785 | 47327
    Dabigatran vs VKA (matched pop): number analyzed (Participants) | 20489 | 0 | 20489 | 40978
    Dabigatran vs VKA (matched pop): Male | 11164 |  | 11164 | 22328
    Dabigatran vs VKA (matched pop): Female | 9325 |  | 9325 | 18650
    Rivaroxaban vs VKA (matched pop): number analyzed (Participants) | 0 | 23053 | 23053 | 46106
    Rivaroxaban vs VKA (matched pop): Male |  | 12557 | 12557 | 25114
    Rivaroxaban vs VKA (matched pop): Female |  | 10496 | 10496 | 20992

OUTCOME MEASURES:

1. Primary Outcome: Clinically Relevant Bleeding
Description: First hospitalization with primary diagnosis (Tenth Revision codes of the International Classification of Diseases (ICD-10 codes)) of:
  1. Hemorrhagic stroke,
  2. Other critical organ or site bleeding,
  3. Other bleeding (gastro-intestinal bleeding, urogenital bleeding and other bleeding subtype).
Time Frame: One year
Population: Patients (pts) with a first dispensing (dispen.) of DOAC or VKA in 2013 for NVAF. For each comparison (dabigatran versus VKA and rivaroxaban versus VKA), patients were matched 1:1 on the date of the first drug (DOAC or VKA) dispensing (± 2 weeks (wks.)), gender, age at index date (± 1 year (yr)) and high-dimensional propensity score (hdPS, ± 0.05).
Measure: Number; unit: participants with event
Groups:
- Dabigatran (Dabigatran vs VKA): Patients with a first dispensing of dabigatran in 2013 for NVAF, matched 1:1 on the date of the first dispensing, gender, age at index date, and hdPS.
- VKA (Dabigatran vs VKA); VKA (Rivaroxaban vs VKA): Patients with a first dispensing of VKA in 2013 for NVAF, matched 1:1 on the date of the first dispensing, gender, age at index date, and hdPS.
- Rivaroxaban (Rivaroxaban vs VKA): Patients with a first dispensing of rivaroxaban in 2013 for NVAF, matched 1:1 on the date of the first dispensing, gender, age at index date, and hdPS.
Arm/Group | Dabigatran (Dabigatran vs VKA) | VKA (Dabigatran vs VKA) | Rivaroxaban (Rivaroxaban vs VKA) | VKA (Rivaroxaban vs VKA)
Number analyzed (Participants) | 20489 | 20489 | 23053 | 23053
participants with event | 367 [2.2 to 2.7] | 668 [4.1 to 4.8] | 635 [3.5 to 4.1] | 767 [4.2 to 4.8]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs VKA) vs VKA (Dabigatran vs VKA); Outcome was analyzed during dabigatran or VKA exposure period (on treatment) using: 1) Cumulative function to estimate the incidence (with death as a competing risk), 2) Fine and Gray model to compare the 1-year risk for dabigatran versus VKA, with hazard ratio (HR) and 95% Confidence Interval (CI ) (and death as a competing risk); Test type: Superiority or Other; p < 0.0001, Fine and Gray model; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.51 to 0.66]
Statistical Analysis 2: Comparison: Rivaroxaban (Rivaroxaban vs VKA) vs VKA (Rivaroxaban vs VKA); Outcome was analyzed during rivaroxaban or VKA exposure period (on treatment) using: 1) Cumulative function to estimate the incidence (with death as a competing risk), 2) Fine and Gray model to compare the 1-year risk for rivaroxaban versus VKA, with HR and 95%CI (and death as a competing risk); Test type: Superiority or Other; p = 0.0006, Fine and Gray model; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.75 to 0.92]

2. Primary Outcome: Major Bleeding
Description: First hospitalization with primary diagnosis (ICD-10 codes) of:
  1. Hemorrhagic stroke,
  2. Other critical organ or site bleeding,
  3. Other bleeding with transfusion, or acute post-hemorrhagic anemia or death during hospital stay.
Time Frame: 1 year
Population: Patients with a first dispensing of DOAC or VKA in 2013 for NVAF. For each comparison (dabigatran versus VKA and rivaroxaban versus VKA), patients were matched 1:1 on the date of the first drug (DOAC or VKA) dispensing (± 2 weeks), gender, age at index date (± 1 year) and high-dimensional propensity score (hdPS, ± 0.05).
Measure: Number; unit: participants with events
Arm/Group | Dabigatran (Dabigatran vs VKA) | VKA (Dabigatran vs VKA) | Rivaroxaban (Rivaroxaban vs VKA) | VKA (Rivaroxaban vs VKA)
Number analyzed (Participants) | 20489 | 20489 | 23053 | 23053
participants with events | 178 [1.0 to 1.4] | 341 [2.0 to 2.5] | 280 [1.5 to 1.9] | 417 [2.2 to 2.7]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs VKA) vs VKA (Dabigatran vs VKA); Outcome was analyzed during dabigatran or VKA exposure period (on treatment) using: 1) Cumulative function to estimate the incidence (with death as a competing risk), 2) Fine and Gray model to compare the 1-year risk for dabigatran versus VKA, with hazard ratio (HR) and 95%CI (and death as a competing risk); Test type: Superiority or Other; p < 0.0001, Fine and Gray model; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.46 to 0.66]
Statistical Analysis 2: Comparison: Rivaroxaban (Rivaroxaban vs VKA) vs VKA (Rivaroxaban vs VKA); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Fine and Gray model; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.58 to 0.79]

3. Primary Outcome: Arterial Thrombotic Event
Description: First hospitalization with primary diagnosis (ICD-10 codes) of:
  1. Ischemic or undefined stroke,
  2. Systemic arterial embolism.
Time Frame: 1 year
Population: as for outcome 2
Measure: Number; unit: participants with events
Arm/Group | Dabigatran (Dabigatran vs VKA) | VKA (Dabigatran vs VKA) | Rivaroxaban (Rivaroxaban vs VKA) | VKA (Rivaroxaban vs VKA)
Number analyzed (Participants) | 20489 | 20489 | 23053 | 23053
participants with events | 226 [1.4 to 1.8] | 321 [1.9 to 2.4] | 343 [1.8 to 2.2] | 351 [1.9 to 2.3]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs VKA) vs VKA (Dabigatran vs VKA); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0007, Fine and Gray model; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.63 to 0.88]
Statistical Analysis 2: Comparison: Rivaroxaban (Rivaroxaban vs VKA) vs VKA (Rivaroxaban vs VKA); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8341, Fine and Gray model; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.85 to 1.14]

4. Primary Outcome: Acute Coronary Syndrome
Description: First hospitalization with primary diagnosis (ICD-10 codes) of:
  1. Myocardial infarction (ST-segment elevation Myocardial infarction (STEMI) and non-ST-segment elevation Myocardial infarction(NSTEMI)),
  2. Unstable angina.
Time Frame: One year
Population: as for outcome 2
Measure: Number; unit: participants with events
Arm/Group | Dabigatran (Dabigatran vs VKA) | VKA (Dabigatran vs VKA) | Rivaroxaban (Rivaroxaban vs VKA) | VKA (Rivaroxaban vs VKA)
Number analyzed (Participants) | 20489 | 20489 | 23053 | 23053
participants with events | 176 [1.1 to 1.4] | 238 [1.4 to 1.8] | 230 [1.2 to 1.5] | 277 [1.4 to 1.8]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs VKA) vs VKA (Dabigatran vs VKA); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0147, Fine and Gray model; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.95]
Statistical Analysis 2: Comparison: Rivaroxaban (Rivaroxaban vs VKA) vs VKA (Rivaroxaban vs VKA); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0501, Fine and Gray model; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 1.00]

5. Primary Outcome: Death (All-cause)
Description: All-cause death (cause of death not available in the database).
Time Frame: 1 year
Population: as for outcome 2
Measure: Number; unit: participants with events
Arm/Group | Dabigatran (Dabigatran vs VKA) | VKA (Dabigatran vs VKA) | Rivaroxaban (Rivaroxaban vs VKA) | VKA (Rivaroxaban vs VKA)
Number analyzed (Participants) | 20489 | 20489 | 23053 | 23053
participants with events | 686 [4.6 to 5.3] | 983 [6.4 to 7.3] | 908 [5.2 to 6.0] | 1186 [6.9 to 7.8]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs VKA) vs VKA (Dabigatran vs VKA); Outcome was analyzed during dabigatran or VKA exposure period (on treatment) using: 1) Kaplan-Meier to estimate the cumulative incidence, 2) Cox proportional hazard risk model to compare the 1-year risk for dabigatran versus VKA, with HR and 95%CI; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard risk model; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.67 to 0.82]
Statistical Analysis 2: Comparison: Rivaroxaban (Rivaroxaban vs VKA) vs VKA (Rivaroxaban vs VKA); Outcome was analyzed during rivaroxaban or VKA exposure period (on treatment) using: 1) Kaplan-Meier to estimate the cumulative incidence, 2) Cox proportional hazard risk model to compare the 1-year risk for rivaroxaban versus VKA, with HR and 95%CI; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard risk model; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.71 to 0.84]

6. Primary Outcome: Composite Criterion (Clinically Relevant Bleeding, Arterial Thrombotic Events, Acute Coronary Syndrome, Death)
Description: First event among clinically relevant bleeding, arterial thrombotic event, acute coronary syndrome, or death defined above.
Time Frame: One year
Population: as for outcome 2
Measure: Number; unit: participants with events
Arm/Group | Dabigatran (Dabigatran vs VKA) | VKA (Dabigatran vs VKA) | Rivaroxaban (Rivaroxaban vs VKA) | VKA (Rivaroxaban vs VKA)
Number analyzed (Participants) | 20489 | 20489 | 23053 | 23053
participants with events | 1340 [8.8 to 9.8] | 1970 [12.5 to 13.7] | 1967 [11.1 to 12.1] | 2328 [13.2 to 14.3]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs VKA) vs VKA (Dabigatran vs VKA); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard risk model; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.66 to 0.76]
Statistical Analysis 2: Comparison: Rivaroxaban (Rivaroxaban vs VKA) vs VKA (Rivaroxaban vs VKA); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard risk model; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.79 to 0.89]

ADVERSE EVENTS:
Description: Claims and hospitalization database without any adverse event declaration, and using secondary individual anonymous information. Thus all outcomes studied were reported in aggregate in the final study report.
Arm/Group | Dabigatran | Rivaroxaban | Vitamin K Antagonists
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
DOAC & VKA were prescribed by physicians in their daily practice,with differences for pts & disease characteristics,including stroke & bleeding risk factors.To control this pts were 1:1 matched on date of 1st dispensing, gender,age & hdPS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.